CLINICAL TRIAL: NCT06359717
Title: Prostatic Specific Membrane Antigen Reporting and Data System (PSMA-RADS) Version 1.0: Prospective Validation and Comparison to Updated Version (v2.0)
Brief Title: Prospective Validation of PSMA-RADS
Acronym: PSMA-RADS
Status: Active, not recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohammad Abd Alkhalik Basha, Principal Investigator, Zagazig University
Other Study IDs: ZU-10490
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cancer Prostate
Keywords: gallium 68 PSMA-11; Prostatic Neoplasms; Positron Emission Tomography; Computed Tomography; Prospective Studies
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 164 new diagnoses, 108 BCR, and 171 follow-up: 1. 164 new diagnoses. 2.108 BCR. 3. 171 follow-up

SUMMARY:
This is a prospective, multicenter study aimed at evaluating the diagnostic accuracy and reliability of the Prostate-Specific Membrane Antigen Reporting and Data System (PSMA-RADS) version 1.0 in detecting prostate cancer using 68Ga-PSMA-11 PET/CT imaging. The study also compared the performance of PSMA-RADS v1.0 with the updated version 2.0.

Key points:

* 477 patients with newly diagnosed, recurrent or follow up prostate cancer underwent 68Ga-PSMA-11 PET/CT imaging.
* Three radiologists independently evaluated the scans and assigned PSMA-RADS scores using v1.0, then retrospectively using v2.0.
* Diagnostic accuracy was assessed against histopathology and follow-up imaging as reference standards.
* Inter-rater agreement was evaluated using Fleiss' kappa statistic.
* The study aimed to validate the diagnostic utility of PSMA-RADS v1.0 and compare it to the updated v2.0.

DETAILED DESCRIPTION:
Study Design and Patient Population:

Between January 2023 and August 2024, a total of 477 consecutive patients were recruited from four institutions. The study cohort included patients with newly diagnosed Pca referred for initial staging, patients with biochemical recurrence (BCR), and patients referred for follow-up. Patients were excluded based on the following criteria: inability to undergo PET/CT scan due to weight (e.g., >180 kg) (n= 4), claustrophobia or inability to lie still throughout the scanning duration (n= 6), allergy to contrast media (n= 3), hepatic impairment (n= 9), renal failure (n= 3), and patients lost during follow-up (n= 9). This resulted in a final cohort of 443 patients (164 new diagnoses, 108 BCR, and 171 follow-up). The flowchart of the study is illustrated in Fig. 1. Once enrolled; all patients underwent a 68Ga-PSMA-11 PET/CT scan. For each patient, we determined the prostate-specific antigen (PSA) value, Gleason score (GS), and disease stage according to the TNM classification (molecular imaging TM (miTNM)), as proposed by PROMISE criteria.

Imaging Protocol:

* All patients underwent 68Ga-PSMA-11 PET/CT imaging on integrated PET/CT scanners.
* Detailed acquisition protocol is provided, including patient preparation, radiotracer dosing, low-dose CT, PET acquisition, and diagnostic contrast-enhanced CT.

Image Analysis:

* Three experienced nuclear medicine radiologists independently evaluated the anonymized PET/CT images in random order, blinded to clinical data.
* They underwent standardized training on PSMA-RADS criteria before the study.
* For each patient, the scan was divided into 4 regions: prostate/bed, lymph nodes, bones, soft tissues.
* Each region was assessed for uptake intensity, sites relevant for metastases, and CT lesion definition.
* Radiologists assigned PSMA-RADS categories (1-5) to each region and an overall patient score using v1.0 criteria.
* Retrospectively, they re-assigned scores using the updated PSMA-RADS v2.0 criteria after its publication in July 2023.

Reference Standard:

The primary endpoint was diagnostic accuracy on a per-patient basis. For newly diagnosed patients (n= 167), the definitive diagnosis was validated by histopathological results after biopsy. Biopsies were obtained through a transrectal ultrasound (TRUS) guided procedure within two weeks before 68Ga-PSMA-11 PET/CT imaging. For patients with biochemical recurrence, and patients with follow-up, the final diagnosis was confirmed based on the following: (i) Histopathological findings after biopsy (n= 151 patients (55 locoregional, 96 lymph nodes, 45 bone lesions, and 42 visceral soft tissue lesions)). Biopsies were taken by ultrasound-guided (n=78) or CT-guided (n=73) procedure within two weeks before 68Ga-PSMA-11 PET/CT imaging. Two experienced pathologists evaluated all specimens, and the results were obtained by consensus. In patients with multiple lesions, the biopsy result of one lesion was considered representative of all lesions. Biopsies were performed to determine the lesion type as per the doctor's request. (ii) One year of clinical and imaging follow-up (n= 37). Follow-up imaging was completed every six months via 68Ga-PSMA-11 PET/CT analysis. It was interpreted by a panel of expert readers who were informed of the locations of the lesions described by the blinded readers at initial imaging.

Statistical Analysis:

* Diagnostic accuracy was evaluated using a 4-fold table against the reference standard.
* ROC analysis was performed to determine optimal cut-offs and AUCs.
* Inter-rater agreement was assessed using Fleiss' kappa statistic.
* Performance of PSMA-RADS v1.0 and v2.0 were compared.

In summary, this prospective study rigorously evaluated the diagnostic performance and reliability of PSMA-RADS v1.0 on a multi-center cohort using 68Ga-PSMA-11 PET/CT, and compared it head-to-head with the updated version 2.0, with thorough statistical analyses planned.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed prostate cancer
2. Patients with biochemical recurrence of prostate cancer
3. Ability to undergo 68Ga-PSMA-11 PET/CT imaging (e.g., no contraindications such as weight limitations, claustrophobia, inability to lie still)
4. No allergy to contrast media used for the diagnostic CT component
5. Adequate hepatic and renal function to receive the radiotracer
6. Willingness to provide informed consent for participation in the study

Exclusion Criteria:

1. Inability to undergo PET/CT scan due to weight (e.g., >180 kg) (n=5)
2. Claustrophobia or inability to lie still throughout the scanning duration (n=3)
3. Allergy to contrast media (n=2)
4. Hepatic impairment (n=5)
5. Renal failure (n=2)
6. Patients lost during follow-up (n=7)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: * A total of 477 consecutive patients were initially recruited from three institutions between January 2023 and August 2024.
  * After applying the exclusion criteria, the final study cohort comprised 443 patients.
  * The cohort included three groups of patients:
    164 new diagnoses, 108 BCR, and 171 follow-up
Sampling Method: Non-Probability Sample
Enrollment: 477 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of PSMA-RADS v1.0 and v2.0 | One year
  The diagnostic accuracy of PSMA-RADS version 1.0 and version 2.0 for detecting prostate cancer lesions using 68Ga-PSMA-11 PET/CT. Diagnostic accuracy will be evaluated using sensitivity, specificity, positive predictive value, and negative predictive value, calculated on a per-patient basis. Histopathological results from biopsy and/or clinical/imaging follow-up will serve as the reference standard

SECONDARY OUTCOMES:
Inter-rater Agreement of PSMA-RADS v1.0 and v2.0 | One year
  The degree of agreement among the three nuclear medicine radiologists in assigning PSMA-RADS categories using version 1.0 and version 2.0 criteria. Inter-rater agreement will be evaluated using Fleiss' kappa statistics

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A. Basha, MD, Principal Investigator — Zagazig University
Locations (1):
- Mohammad Abd Alkhalik Basha, Zagazig, Select, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT06359717/Prot_SAP_000.pdf